CLINICAL TRIAL: NCT00828659
Title: A Randomized, Double-Blind, Double-Dummy, Placebo- and Active-Controlled Crossover Study to Evaluate the Abuse Potential of Single Doses of Lorcaserin in Healthy Recreational Polydrug Users
Brief Title: Abuse Potential of Single Doses of Lorcaserin in Healthy Recreational Polydrug Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: APD356-013
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2009-07

CONDITIONS: Drug Abuse; Healthy
Keywords: Abuse potential
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Active Comparator #1 (Active Comparator)
  Interventions: Drug: Active Comparator #1
- Active Comparator #2 (Active Comparator)
  Interventions: Drug: Active Comparator #2
- Active Comparator #3 (Active Comparator)
  Interventions: Drug: Active Comparator #3
- Lorcaserin Dose #1 (Experimental)
  Interventions: Drug: Lorcaserin Dose #1
- Lorcaserin Dose #2 (Experimental)
  Interventions: Drug: Lorcaserin Dose #2
- Lorcaserin Dose #3 (Experimental)
  Interventions: Drug: Lorcaserin Dose #3

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Active Comparator #1
  Arms: Active Comparator #1
Drug: Active Comparator #2
  Arms: Active Comparator #2
Drug: Active Comparator #3
  Arms: Active Comparator #3
Drug: Lorcaserin Dose #1
  Arms: Lorcaserin Dose #1
Drug: Lorcaserin Dose #2
  Arms: Lorcaserin Dose #2
Drug: Lorcaserin Dose #3
  Arms: Lorcaserin Dose #3

SUMMARY:
The purpose of this study is to evaluate the abuse potential of lorcaserin in healthy recreational polydrug users.

ELIGIBILITY:
INCLUSION CRITERIA

1. Healthy male or female subjects 18 to 55 years of age, inclusive.
2. Body mass index (BMI) within the range of 18 to 33 kg/m2, inclusive, and a minimum weight of at least 50 kg at Screening.
3. Free from any clinically significant medical or psychiatric abnormality
4. Recreational polydrug user with a history of psychedelic and depressant drug use,and at least one occasion of use in the past 3 months.
5. Female subjects must have a negative serum pregnancy test at Screening and urine pregnancy test at each admission.
6. Female subjects of childbearing potential must be practising abstinence or using and willing to continue using a medically acceptable form of birth control for at least 1 month after the last study drug administration. Male subjects who have female partners of childbearing potential must ensure that their partner use an acceptable method of contraception.
7. Willingness to take a drug that might alter perception in a controlled setting.

EXCLUSION CRITERIA

A subject will not be considered eligible to participate in this study, if any one of the following exclusion criteria is satisfied:

1. A history or presence of drug or alcohol dependence (excluding nicotine and caffeine).
2. Use of non-prescription, prescription medication or natural health products (except acetaminophen, vitamin or mineral supplements, acceptable forms of birth control, and hormone replacement) within 7 days prior to first drug administration in the qualification phase and throughout the study.
3. Use of SSRIs (e.g. fluoxetine, paroxetine, citalopram) within 14 days prior to first drug administration in the qualification phase and throughout the study.
4. History of allergy or hypersensitivity to the study drugs
5. Female subjects who are currently pregnant or lactating or who are planning to become pregnant within 30 days of last study drug administration
6. Treatment with any investigational drug within 30 days prior to first drug administration during the qualification phase.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the abuse potential of lorcaserin

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of lorcaserin

CONTACTS AND LOCATIONS:
Locations (1):
- Kendle Early Phase, Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Shram MJ, Schoedel KA, Bartlett C, Shazer RL, Anderson CM, Sellers EM. Evaluation of the abuse potential of lorcaserin, a serotonin 2C (5-HT2C) receptor agonist, in recreational polydrug users. Clin Pharmacol Ther. 2011 May;89(5):683-92. doi: 10.1038/clpt.2011.20. Epub 2011 Mar 16. PMID 21412231